CLINICAL TRIAL: NCT01868789
Title: In-Vivo Physiologic Weight-Bearing Assessment of Tarsal Instability: Three-Dimensional Cone-Beam Computed Tomography Analysis
Brief Title: Weightbearing Assessment of Tarsal Instability
Acronym: WBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedic Foot and Ankle Center, Ohio (Other)
Collaborators: CurveBeam LLC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OH1-12-00397
Record Dates: First submitted 2013-05-24; First posted 2013-06-05 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Adult-acquired Flatfoot Disorder (AAFD)
Keywords: Adult-acquired flatfoot disorder (AAFD); flexible flatfoot; computed tomography (CT)
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weightbearing CT (AAFD group) (Experimental): Weightbearing CT scan of affected foot
  Interventions: Radiation: Weightbearing CT
- Weightbearing CT (control group) (Active Comparator): Weightbearing CT scan of normal foot
  Interventions: Radiation: Weightbearing CT

INTERVENTIONS:
Radiation: Weightbearing CT

SUMMARY:
The purpose of this study is to compare the average joint motion and joint axis orientation of the hindfoot bones between patients diagnosed with adult-acquired flatfoot disorder (AAFD) and a control group of patients without foot deformity, using weight-bearing CT technology.

ELIGIBILITY:
Symptomatic group:

Inclusion Criteria:

1. adult patients (ages 18 -80 years old) diagnosed with Stage 2 AAFD

Exclusion Criteria:

1. previous surgery
2. infection
3. tumor in the affected foot
4. pregnancy

Control group:

Inclusion Criteria:

1. adult patients (ages 18 -80 years old) without foot deformity

Exclusion Criteria:

1. history of previous foot and ankle surgery
2. foot deformity
3. known foot and ankle pathology
4. pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Berlet, MD, Principal Investigator — Orthopedic Foot and Ankle Center
Locations (1):
- Orthopedic Foot and Ankle Center, Westerville, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Weightbearing CT (AAFD Group): Weightbearing CT scan of affected foot
  Weightbearing CT
- Weightbearing CT (Control Group): Weightbearing CT scan of normal foot
  Weightbearing CT
Period: Overall Study
Arm/Group | Weightbearing CT (AAFD Group) | Weightbearing CT (Control Group)
Started | 9 | 14
Completed | 7 | 12
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weightbearing CT (AAFD Group) | Weightbearing CT (Control Group) | Total
Number analyzed (Participants) | 7 | 12 | 19
Age, Continuous [Mean (Full Range); unit: years] | 43.6 [19.6 to 69.3] | 52.2 [30.6 to 82.0] | 49.0 [19.6 to 82.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Joint Motion Between Touch-down Bearing Navicular and Full-weight Bearing Navicular
Description: Relative motion, which is the position of the full weightbearing (FWB, greater that 75-100% body weight) navicular in comparison to the touch down weightbearing (TDWB, 25-50% body weight) navicular position, will be determined by comparing the joint orientation across these two points on one CT scan. The difference between the two positions is reported below.
Time Frame: 1 CT scan, one reading while touch-down bearing, one reading while full-weight bearing
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Weightbearing CT (AAFD Group) | Weightbearing CT (Control Group)
Number analyzed (Participants) | 7 | 12
mm
  Translation of the Navicular | 3.56 (2.15) | 4.36 (2.16)
  axis of navicular rotation: x component | -0.1666 (0.338) | -0.170 (0.188)
  axis of navicular rotation: y component | 0.867 (0.159) | 0.950 (0.045)
  axis of navicular rotation: z component | -0.083 (0.331) | 0.084 (0.171)

2. Primary Outcome: Change in Navicular Rotation Between Touch-down Bearing and Full-weight Bearing
Description: Relative motion across joint segments will be determined by comparing the joint orientation across two time points: touch-down bearing (TDWB, 25-50% body weight) and full-weight bearing (FWB, greater that 75-100% body weight) as measured on CT.
Time Frame: 1 CT scan, one reading while touch-down bearing, one reading while full-weight bearing
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Weightbearing CT (AAFD Group) | Weightbearing CT (Control Group)
Number analyzed (Participants) | 7 | 12
degrees | 4.11 (2.19) | 5.99 (3.26)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Weightbearing CT (AAFD Group) | Weightbearing CT (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 0/9 | 0/13

LIMITATIONS AND CAVEATS:
Any movement during the scanning process or metal implants caused difficulty with reconstructing the positioning of the bones, therefore those subjects were eliminated from analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes